CLINICAL TRIAL: NCT04635007
Title: The Effect of Pre-operative Intravenous Tranexamic Acid Versus Rectal Misoprostol in Reducing Blood Loss During and After Elective Cesarean Section in Primigravida: A Double-blinded, Randomized, Controlled Trial
Brief Title: Tranexamic Acid Versus Misoprostol in Reducing Blood Loss in Cesarean Section in Primigravida
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AN2020
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Cesarean Section Complications; Blood Loss, Surgical; Misoprostol; Tranexamic Acid
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Misoprostol

STUDY DESIGN:
Intervention Model Description: The patients will be divided into 2 groups
  Group no. (1) 100 women: will receive preoperative 1 gram of TXA (kapron®, Amoun, Egypt) 10 minutes before skin incision, by slow intravenous injection over 10 minutes (Tranexamic acid injection will be prepared by diluting 1gm (10ml) TXA in 100 ml. of normal saline. TXA will be administrated as an intravenous infusion or slowly injection) and preoperative placebo (4 tablets similar to misoprostol in size and shape as peroxide) will be administrated rectally.
  Group no. (2) 100 women: will receive preoperative 800 micrograms of misoprostol (4 tablets) rectally after spinal anesthesia and urinary catheterization (as per WHO dose recommendation) (Conde-Agudelo et al., 2013) and preoperative placebo (10 minutes before skin incision, 10 ml of distilled water ampoules by slow intravenous injection over 10 minutes).
Who Masked: Participant, Investigator
Masking Description: A double-blind study is one in which neither the participants nor the experimenters know who is receiving a particular treatment. This procedure is utilized to prevent bias in research results. Double-blind studies are particularly useful for preventing bias due to demand characteristics or the placebo effect. In a double-blind study, the investigators who interact with the participants would not know who will receive the actual drug and who will receive a placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Tranexamic acid group (Experimental): 100 women: will receive preoperative 1 gram of TXA (kapron®, Amoun, Egypt) 10 minutes before skin incision, by slow intravenous injection over 10 minutes (Tranexamic acid injection will be prepared by diluting 1gm (10ml) TXA in 100 ml. of normal saline. TXA will be administrated as an intravenous infusion or slowly injection) and preoperative placebo (4 tablets similar to misoprostol in size and shape as peroxide) will be administrated rectally.
  Interventions: Drug: Tranexamic acid
- Group 2: Misoprostol group (Experimental): 100 women: will receive preoperative 800 micrograms of misoprostol (4 tablets) rectally after spinal anesthesia and urinary catheterization (as per WHO dose recommendation) (Conde-Agudelo et al., 2013) and preoperative placebo (10 minutes before skin incision, 10 ml of distilled water ampoules by slow intravenous injection over 10 minutes).
  Interventions: Drug: Misoprostol 200mcg Tab

INTERVENTIONS:
Drug: Tranexamic acid — 100 women: will receive preoperative 1 gram of TXA (kapron®, Amoun, Egypt) 10 minutes before skin incision, by slow intravenous injection over 10 minutes (Tranexamic acid injection will be prepared by diluting 1gm (10ml) TXA in 100 ml. of normal saline. TXA will be administrated as an intravenous infusion or slowly injection) and preoperative placebo (4 tablets similar to misoprostol in size and shape as peroxide) will be administrated rectally.
  Other Names: Kapron
  Arms: Group 1: Tranexamic acid group
Drug: Misoprostol 200mcg Tab — 100 women: will receive preoperative 800 micrograms of misoprostol (4 tablets) rectally after spinal anesthesia and urinary catheterization (as per WHO dose recommendation) (Conde-Agudelo et al., 2013) and preoperative placebo (10 minutes before skin incision, 10 ml of distilled water ampoules by slow intravenous injection over 10 minutes).
  Other Names: Cytotic
  Arms: Group 2: Misoprostol group

SUMMARY:
The aim of the work is to compare the efficacy of preoperative IV tranexamic acid and rectal misoprostol in reducing blood loss in the elective cesarean section.

Research question:

In women undergoing elective cesarean section, is preoperative administration of IV tranexamic acid better than rectal misoprostol in reducing blood loss?

DETAILED DESCRIPTION:
* Type of study: Prospective double-blinded randomized placebo-controlled Clinical trial
* Time plan: Approximately 12 months according to calculated sample size.
* study setting: this study will be conducted obstetrics and gynecology department at Cairo University.
* study population: Patients will be enrolled in this study of those attending the obstetric clinic at kasr el ainy hospital for elective cesarean section.
* Methodology:

  * Methodology in details:
  * Verbal and written consent will be obtained before history taking All women will be subjected to

History taking:

* Detailed clinical history.
* Personal history:

Name, Age, Parity, Occupation, Residency, and Special habits.

-Present history: History of onset, course, and duration of vaginal bleeding or bloody vaginal discharge, presence of uterine contraction, PROM, IUGR, or any indication for cesarean section.

-Obstetric history: History of previous abortion.

-Menstrual history: For estimation of gestational age using Naegele's rule, provided that she had regular cycles for the last three months before she got pregnant and was not taking contraceptive pills during this period and she was sure of her dates.

Term pregnancy defined as delivery between 37 and 42 weeks of gestation. Gestational age will be assessed from the menstrual history and will be confirmed by measurement of fetal crown-rump length at a first-trimester scan.

-Past history: History of medical disorders, drug therapy or allergy, or history of intake of other tocolytic drugs.

-Family history: For consanguinity in the case of CFMF.

Examination

* Full clinical examination (pulse, temperature, and blood pressure).
* General examination including blood pressure, heart rate, body temperature, body mass index, head& neck examination, Bilateral lower limb examination, chest, heart.
* Local clinical examination; assessment of maternal health, obstetric abdominal examination for fundal level, fetal presentation, estimating fetal weight, and scars of previous operations, uterine contraction if present, auscultation of FHR.
* Preoperative investigations (Rh, CBC, HTC, Hb, Coagulation profile, fasting and postprandial blood sugar, and complete urine analysis).
* Ultrasonography examination: to assess the following data:
* Gestational age
* Fetal viability
* Fetal presentation and EFW.
* Detection of any fetal congenital anomalies.
* To ensure that all inclusion criteria are present.
* Check amniotic fluid index (the amniotic fluid index (AFI) will be estimated using abdominal ultrasonography on the day of delivery or the day before delivery. The uterus will be divided into four quadrants; the right and left quadrants will be defined by the linea nigra, and the upper and lower quadrants will be defined by the umbilicus. The maximum vertical diameter of amniotic fluid in each quadrant will be measured in centimeters. The sum of these four quadrants will be used to calculate the AFI. The volume of amniotic fluid in ml. will be estimated by multiplying the AFI by 30.

Intervention:

The cesarean section will be done by a senior registrar who performed at least 300 cesarean sections before the start of the study. All CS will be performed using spinal anesthesia; the abdomen will be entered by Pfannenstiel abdominal incision.

The allotted sealed envelope (allocation concealment will be discussed later) will be taken to the theatre and handed over to the anesthetist who will administrate the drug (TXA or Misoprostol) or the placebo to the patient without telling neither the researcher nor the patient the content of the envelope. With the induction of anesthesia, patients assigned to group 1 will receive 1 gram of TXA (kapron®, Amoun, Egypt) 10 minutes before skin incision, by slow intravenous injection over 10 minutes and preoperative placebo (4 tablets similar to misoprostol in size and shape as peroxide) will be administrated rectally. (Tranexamic acid injection will be prepared by diluting 1gm (10ml) TXA in 100 ml of normal saline. Participants are assigned to group 2 will receive 800μg rectal misoprostol (Misotac®, SIGMA, Egypt) immediately after urinary catheterization and before skin incision and preoperative placebo (10 minutes before skin incision, 10 ml of distilled water ampoules or normal saline by slow intravenous injection over 10 minutes).

All women will receive 10 IU of oxytocin (syntocinon®, NOVARTIS) by slow intravenous after cord clamping.

Sterilization and toweling of the patient then the standard technique of trans-peritoneal lower segment cesarean will be adopted. The placenta will be removed by cord traction and uterine compression. The uterus will be exteriorized and compressed during closure which will be achieved by continuous unlocked sutures in 2 layers using 2/0 polyglactin suture and 1 cm interval between sutures. The peritoneum and muscle will be closed by 2/0 polyglactin suture and the sheath will be closed by 1/0 polyglactin, and the skin will be closed by subcuticular suture using proline double zero suture in both groups. The estimation of blood loss will be started after skin incision.

* The linen towels will be weighted in (mg) with its cover before and after the operation using a highly accurate digital balance and the difference in weight between dry and soaked linen towels will be calculated.
* Blood loss during the operation will be calculated as follows:
* Volume of the contents of the suction bottle (ml) (A).
* Difference in weight of linen towels (gm) (B) (weight of soaked linen towels (gm) - the weight of dry linen towels (gm)).
* Amniotic fluid volume (ml) (C).
* So, blood loss during operation (ml) = (A + B) - C.
* Allowable blood loss will be calculated for all women according to the underlying law.

ABL= EBV x (Hi - Hf) / Hi

Hi = initial Hct Hf = final lowest acceptable Hct Estimated Blood Volume (EBV) EBV = weight (kg) X average blood volume (75-85 ml/kg)

* A trained nurse will be responsible for the collection of wound dressing placed in the vulval area during the first 24 hours after surgery and the difference in weight will be calculated. The overall blood loss will be calculated.
* The difference between preoperative and 24 hours postoperative in hemoglobin concentration and hematocrit value will be measured to calculate allowable blood loss
* The need for additional uterotonics drugs will be given according to the attendant consultant decision or a blood loss of more than 1000ml intraoperative.
* Operative time, need for blood transfusion and side effects of study drug e.g. nausea, vomiting, diarrhea will be recorded.
* All the patients will receive non-steroidal anti-inflammatory preparation in the form of (Rheumarene®) 75mg IM (one ampoule) immediately postoperative than one ampoule 12 hours postoperative and the need for extra analgesics will be recorded.
* All the patients will receive prophylactic broad-spectrum antibiotics in form of (Ceftriaxone®, Sandoz, Egypt) 1 gm./12 hours.
* The Apgar score of the fetus at 1 and 5 minutes, the need for neonatal intensive care unit (NICU) admission, and neonatal death will be assessed in the two groups.
* Data will be collected, tabulated, and statistically analyzed by IBM computer using the Statistical Package for the Social Sciences (SPSS version 24). Chi-square test will be used to compare qualitative variables between groups and Fisher exact test will be used instead of the Chi-square test when the expected cell count less than 5. The student t-test will be used to compare the quantitative variables in parametric data. P-value <0.05 will be set signiﬁcant.

ELIGIBILITY:
Inclusion Criteria:

* Women booked for a primary elective cesarean section, not in active labor
* Aged between 18-40 years.
* BMI 18.5-29.9 kg/ m2 pre-pregnancy weight
* Term pregnancies (Early term: between 37 weeks, 0 days and 38 weeks, 6 days. Full term: between 39 weeks, 0 days and 40 weeks, 6 days. Late term: between 41 weeks, 0 days and 41 weeks, 6 days).
* Singleton pregnancies.
* Indication of elective cesarean section (Malpresentation, Malposition, Cephalopelvic disproportion, active herpes)
* Fetal macrosomia (Macrosomia is defined as birth-weight over 4,000 g irrespective of gestational age)
* Certain congenital fetal malformation and skeletal disorders (Several congenital anomalies are controversial indications for cesarean delivery; these include fetal neural tube defects (to avoid sac rupture), particularly defects that are larger than 5-6 cm in diameter as anterior cystic hygroma vascular sacrococcygeal teratoma, giant omphalocele and hydrocephalus with an enlarged biparietal diameter, and some skeletal dysplasia such as type III osteogenesis imperfecta. (Hamrick et al., 2008)

Exclusion Criteria:

* Placenta previa.
* Maternal hypertension and Preeclampsia.
* Diabetes mellitus.
* Severe medical disorder (renal or hepatic).
* Multiple Fibroid uterus.
* Multiple pregnancies.
* Polyhydramnios.
* Previous uterine surgery as myomectomy.
* Contraindication to spinal anesthesia.
* Blood coagulopathy and bleeding disorder.
* Marked maternal anemia (Preoperative hemoglobin <9 gm/dl).
* Contraindications to prostaglandin therapy (e.g. history of severe bronchial asthma or allergy to misoprostol) or TXA

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Blood loss | 6 hours
  Estimation of Intraoperative and postoperative blood loss.

SECONDARY OUTCOMES:
Maternal outcome | 6 hours
  Need of extra utero-tonic drugs
Maternal outcome | 24 hours
  Incidence of postpartum hemorrhage (defined as bleeding >1000 mL during the first 24 hours after the operation)
maternal outcome | 24 hours
  Need for blood transfusion
Maternal outcome | 24 hours
  Post-operative HB & HTC
Maternal outcome | 12 hours
  The incidence of side effects e.g. nausea, vomiting, diarrhea, shivering and headache.
Maternal outcome | 2 hours
  Duration of operation
maternal outcome | 24 hours
  Time of resuming bowel habits

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Taymour, MD, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine - Cairo university, Cairo, Kasr El Ainy, Egypt